CLINICAL TRIAL: NCT02653261
Title: Safety and Efficacy of Intravenous Tranexamic Acid in Reducing Blood Transfusion After Endoscopic Transurethral Resections in Urology: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Safety and Efficacy of Intravenous Tranexamic Acid in Endoscopic Transurethral Resections in Urology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ali JENDOUBI, MD, Assistant Professor, University Tunis El Manar
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: University Tunis El Manar
Record Dates: First submitted 2016-01-03; First posted 2016-01-12 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Hemorrhage
Keywords: tranexamic acid; Transurethral Resection of the Prostate (TURP); Transurethral Resection of a Bladder Tumor (TURBT); Hemorrhage; Blood Transfusion
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): Tranexamic Acid (TXA): bolus of 10 mg/kg thirty minutes before resection followed by infusion of 1 mg/kg/h intraoperatively and for 24 h postoperatively
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): An equal volume of saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid (TXA) is a synthetic analog of serin than reversibly inhibits fibrinolysis by blocking lysine union sites in the plasmin and plasminogen activator molecules. TXA: bolus of 10 mg/kg thirty minutes before resection followed by infusion of 1 mg/kg/h intraoperatively and for 24 h postoperatively
  Other Names: Exacyl
  Arms: Tranexamic Acid
Drug: Placebo — An equal volume of saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Transurethral resection of the prostate (TURP) represents the gold standard in the operative management of benign prostatic hyperplasia (BPH) and the transurethral resection of bladder tumor (TURBT) is the first-line surgical treatment for bladder tumors. One of the most important complications of urological endoscopic resections is intraoperative and postoperative bleeding requiring blood transfusion. Allogeneic blood transfusion is not free of risks, like infection transmission, hemolytic reactions, transfusion-related lung injury, fluid overload, increased costs and hospital length of stay.

Tranexamic acid (TXA) is a synthetic analog of serin than reversibly inhibits fibrinolysis by blocking lysine union sites in the plasmin and plasminogen activator molecules. TXA has been used to reduce blood loss and the need for allogeneic blood transfusion in cardiac surgery and orthopedic surgical procedures but few studies have assessed the efficacy of this antifibrinolytic agent in urological endoscopic procedures.

The investigators designed this double-blind, placebo controlled study evaluate the safety and efficacy of the antifibrinolytic agent tranexamic acid in reducing blood transfusion in patients undergoing endoscopic surgery in urology.

DETAILED DESCRIPTION:
Participants will be randomized into one of two study groups: Group TXA: intravenous tranexamic acid: bolus of 10 mg/kg thirty minutes before resection followed by infusion of 1 mg/kg/h intraoperatively and for 24 h postoperatively. Control Group C: an equal volume of saline. The study drug was prepared by an anesthesiologist not involved in the patient management and data collection. The anesthetic technique will be standardized. Serum hemoglobin was measured before and after surgery. The volume of the irrigation fluid, resected prostate weight and duration of resection were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>/=18)
2. male or female
3. Undergoing elective TURP or TURBT
4. Spinal anesthesia
5. Subject is American Society of Anesthesiologists (ASA) physical status 1 or 2.

Exclusion Criteria:

1. Atrial fibrillation
2. Coronary artery disease treated with drug eluting stent
3. Severe chronic renal failure
4. Congenital or acquired thrombophilia
5. Known or suspected allergy to tranexamic acid.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of red blood cell transfusions | From surgery until 72 hours postoperatively

SECONDARY OUTCOMES:
The difference in preoperative and postoperative hematocrit levels to estimate blood loss. | the first postoperative day
Episodes of acute urinary retention | the first postoperative day
Postoperative bleeding with clot retention | the first postoperative day
Episodes of bladder tamponade requiring evacuation or reintervention | the first postoperative day
Postoperative myocardial ischemia assessed by cardiac troponin I | the first postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Ali JENDOUBI, Principal Investigator — University Tunis El Manar
Locations (1):
- Ali JENDOUBI, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No